CLINICAL TRIAL: NCT02770313
Title: Weekly ONe-Day WatER-only Fasting InterventionaL Trial for Low-Density Lipoprotein Cholesterol Reduction
Acronym: WONDERFUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1050163
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Intermittent Fasting
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent Fasting (Experimental): Water-only Intermittent Fasting
  Interventions: Behavioral: Intermittent Fasting
- Control (No Intervention): ad libitum Usual Diet

INTERVENTIONS:
Behavioral: Intermittent Fasting — Subjects allocated to the fasting arm will undergo a fasting regimen of twice-per-week 24-hour fasting on non-consecutive days during the first 4 weeks of the study, then once-per-week 24-hour fasting during the rest of the study (22 weeks).
  Arms: Intermittent Fasting

SUMMARY:
The goal of this study is to determine how effective repeated fasting over 26 weeks (6 months) is at improving risk parameters that are surrogate endpoints for cardiovascular diseases, metabolic dysregulation and cognitive impairments.

Subjects will be randomized 1:1 to water-only fasting or to their ad libitum usual diet, with randomization performed within strata based on fasting history (≤180 hours or 181-720 hours of total fasting for >12 consecutive hours per episode in the previous two years). Subjects will be assessed at 4, 13 and 26 weeks following randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female, 21-70 years of age,

   * who are not currently taking a statin medication,
   * who have either pre-diabetes (clinical diagnosis, hemoglobin A1c ≥5.6%, or untreated fasting glucose > 100 mg/dL within 6 months of screening) and are not taking medications to control diabetes OR diagnosed, diet-controlled type 2 diabetes but do not require medications to control diabetes OR one or more of the components of the metabolic syndrome measured within 6 months of screening (other than fasting glucose level >100 mg/dL, i.e.: 1. systolic blood pressure ≥130 mmHg, or diastolic ≥85 mmHg, or use of an antihypertensive medication, 2. high-density lipoprotein cholesterol <40 mg/dL for males or <50 mg/dL for females, 3. triglycerides ≥150 mg/dL or use of a non-statin triglyceride-lowering medication (e.g., fibrate, niacin), 4. waist circumference ≥40 inches (102 cm) for males or ≥35 inches (88 cm) for females, or body mass index >25 kg/m2),
   * are 21-39 years of age with LDL-C (measured within six months of screening) of 90-189 mg/dL OR are 40-70 years of age with LDL-C of 90-159 mg/dL OR are 21-70 years of age with LDL-C of 90 mg/dL or greater who have tried statins and stopped due to intolerance to the medications or who have one or more contraindications to statins and thus cannot take them but meet other study inclusion and exclusion criteria.
2. Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.

Exclusion Criteria:

1. Pregnant and/or lactating women and women of child bearing potential who are not using acceptable means of contraception. Women who become pregnant after enrollment in the study will be withdrawn for the health of the mother and baby.
2. Individuals who have fasted more than 15 hours per episode more than once per month during the past two years (i.e., >720 hours over two years), except for those who fast during multiple weeks once per year (e.g., Muslim, Baha'i) who will be allowed to begin participation starting at two weeks after their preferred annual period of fasting ends (e.g., Ramadan or the Baha'i fast) and ending at six months prior to the beginning of the next annual observance, as long as they do not fast routinely outside of the one annual period of fasting.
3. Refusal to drink water while fasting.
4. Prior diagnosis of a chronic disease (i.e., defined as symptomatic coronary artery disease, coronary revascularization, myocardial infarction, unstable angina, stroke, transient ischemic attack, pulmonary embolism, peripheral vascular thromboembolism, chronic kidney disease stage III or higher, chronic obstructive pulmonary disease, immunodeficiency, solid organ transplant, eating disorder, type I diabetes, dementia, traumatic brain injury including post-concussive syndrome, and cancer of any type within the last 5 years other than cancer of the skin excluding melanoma).
5. Pre-diabetics or diabetics on diabetes medication.
6. Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study.
7. Other conditions that in the opinion of the Principal Investigator may increase risk to the subject and/or compromise the quality of the clinical trial.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Change score of low density lipoprotein cholesterol | 26 weeks

SECONDARY OUTCOMES:
Change score for Homeostatic Model Assessment - Insulin Resistance | 26 weeks
Change score for Metabolic Syndrome Score | 26 weeks
Change score for brain-derived neurotrophic factor (BDNF) level | 26 weeks
Change score for the MicroCog test's general cognitive proficiency index score | 26 weeks

OTHER OUTCOMES:
Change score for gut microbiota composition based on 16S rDNA sequencing | 26 weeks
  Change score for gut microbiota composition based on 16S rDNA sequencing among N=30 participants who opt in to this pre-specified substudy.
  Shannon's diversity index will be used because it measures the uncertainty in finding a specific type of microbe from one that is randomly selected from a stool sample. The index ranges from 0 to infinity. A higher value indicates that more diversity in species exists in the stool sample. It is calculated as negative one multiplied by the sum across each species of the proportion of the whole that the species constitutes in the stool multiplied by the natural log of that proportion. The change score will be the value at week 26 minus the value at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Horne, PhD, MPH, Principal Investigator — Intermountain Heart Institute
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horne BD, Anderson JL, May HT, Bair TL, Le VT, Iverson L, Knowlton KU, Muhlestein JB. Insulin resistance reduction, intermittent fasting, and human growth hormone: secondary analysis of a randomized trial. NPJ Metab Health Dis. 2024 Oct 3;2(1):26. doi: 10.1038/s44324-024-00025-2. PMID 40604163
- [Derived] Bartholomew CL, Muhlestein JB, May HT, Le VT, Galenko O, Garrett KD, Brunker C, Hopkins RO, Carlquist JF, Knowlton KU, Anderson JL, Bailey BW, Horne BD. Randomized controlled trial of once-per-week intermittent fasting for health improvement: the WONDERFUL trial. Eur Heart J Open. 2021 Sep 3;1(2):oeab026. doi: 10.1093/ehjopen/oeab026. eCollection 2021 Sep. PMID 35919268
- [Derived] Horne BD, Anderson JL, May HT, Le VT, Galenko O, Drakos SG, Bair TL, Knowlton KU, Muhlestein JB. Intermittent fasting and changes in Galectin-3: A secondary analysis of a randomized controlled trial of disease-free subjects. Nutr Metab Cardiovasc Dis. 2022 Jun;32(6):1538-1548. doi: 10.1016/j.numecd.2022.03.001. Epub 2022 Mar 7. PMID 35361560